CLINICAL TRIAL: NCT06863623
Title: The Effect of Immersive Virtual Reality and Relaxing Videos on Symptom Severity, Distress and Quality of Life in Patients With Lung Cancer Undergoing Chemotherapy
Brief Title: The Effect of Immersive Virtual Reality and Relaxing Videos on Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kadir Baysoy, Research Assitant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA-22070 (Hacettepe Un.); 21-AKD-31 (Registry Identifier: Republic of Turkey Ministry of Health Turkish Medicines and Medical Devices Agency (TİTCK))
Record Dates: First submitted 2024-11-27; First posted 2025-03-07 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer; Chemotherapy Effect; Distress, Emotional; Quality of Life (QOL)
Keywords: cancer; chemotherapy; immersive; virtual reality; lung cancer; quality of life; symptom; side-effect
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Three-Arm Randomised Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group (Experimental): Immersive Virtual Reality Group: Immersive virtual reality will be applied to this group 2 times during chemotherapy infusion (total of 2 chemotherapy cures) to reduce the symptom severity and distress level and improve the quality of life.
  For Immersive Virtual Reality interventions; The Meta Quest 2 device will be used and the virtual scenarios/contents were selected from "Nature Treks" app bought by the researcher.
  (Initially, a total of 6 VR contents and 6 similar videos were created for patients who received cisplatin+etoposide treatment consisting of three sessions of one chemotherapy cure (4 cure, 12 sessions). Due to the limited number of patients and regular attendance to treatment, other similar drug treatments were also included and finally, a total of 2 cures, 2 VR contents and 2 videos were selected and these 2 contents will be used.)
  These:
  1. Walking in the Fores and Similar Video
  2. Sitting on the Beaach and Similar Video
  Interventions: Other: İmmersive Virtaul Reality Applications
- Relaxing Video Group (Experimental): Relaxing Video Group: Participants in this group will watch relaxing videos 2 times for 20 min during chemotherapy infusion (total of 2 chemotherapy cures) to reduce the symptom severity and distress level and improve the quality of life.
  The videos are slideshow-type videos consisting of various images and relaxing music prepared by the researcher. The videos were created by selecting images/sounds similar with the themes/scenarios in the virtual reality application.
  (Initially, a total of 6 VR contents and 6 similar videos were created for patients who received cisplatin+etoposide treatment consisting of three sessions of one chemotherapy cure (4 cure, 12 sessions). Due to the limited number of patients and regular attendance to treatment, other similar drug treatments were also included and finally, a total of 2 cures, 2 VR contents and 2 videos were selected and these 2 contents will be used.) These:Walking in the Fores and Similar Video Sitting on the Beaach and Similar Video
  Interventions: Other: Relaxing Videos
- Control Group (No Intervention): Patients in the control group will receive standard nursing care applied in the chemotherapy unit. Standard nursing care; Training patients on the method of chemotherapy administration, its duration, content, side effects, and coping, preparing the drugs for administration, preparing the patients for treatment, starting the infusion, monitoring the patients during the infusion for side effects, infusion complications, changes in vital signs, etc. Includes applications.

INTERVENTIONS:
Other: İmmersive Virtaul Reality Applications — To apply immersive virtual reality applications (Scenarios)
  Arms: Virtual Reality Group
Other: Relaxing Videos — To watch relaxing videos including pictures and sounds prepared by researcher
  Arms: Relaxing Video Group

SUMMARY:
Lung cancer is one of the types of cancer with a high incidence and mortality rate in the world and in our country. Frequently used protocols in the chemotherapy treatment of lung cancer are the Platine-based drugs. The main side effects of this chemotherapy protocols are nausea, vomiting, neutropenia and fatigue. The side effects of cancer and chemotherapy cause patients to experience distress and their quality of life is adversely affected. Some non-pharmacological methods such as meditation, breathing exercises, and massage can be used to manage the symptoms experienced by patients due to chemotherapy for supportive care. One of these methods is the virtual reality applications. In addition, audio-visual (video) therapy methods are other methods that can be used in the symptom management of these patients. In this study, the effect of interactive/imersive virtual reality intervention and relaxant video intervention on symptom severity, distress level and quality of life of patients diagnosed with lung cancer will be evaluated. Patients will be assigned to 3 groups: virtual reality intervention group (VR), relaxant video application group (RV) and control group (CG) by stratified randomization according to the disease stage and dryg type. During the chemotherapy treatment, the patients will take interactive/immersibe virtual reality (VR group) or relaxant video application (RV group) consisting of nature-themed scenarios. The interventions will be done 2 times and about 20 minutes in the first day of each chemotherapy cycles, in total 2 cycles. The control group will receive routine nursing care. Research data will be collected at different intervals during the chemotherapy course with the Patient Information Form (only once), the Edmonton Symptom Diagnosis Scale, the NCCN Distress Thermometer, the European Cancer Treatment and Organization Committee Quality of Life Scale and the Patient Follow-up Form and will be analyzed with the IBM SPSS v.23 program.

DETAILED DESCRIPTION:
Lung cancer is one of the types of cancer with a high incidence and mortality rate in the world and in our country. Frequently used protocols in the chemotherapy treatment of lung cancer are the Platine-based drugs. The main side effects of this chemotherapy protocols are nausea, vomiting, neutropenia and fatigue. The side effects of cancer and chemotherapy cause patients to experience distress and their quality of life is adversely affected. In addition to pharmacological approaches, some non-pharmacological methods such as meditation, breathing exercises, and massage can be used to manage the symptoms experienced by patients due to chemotherapy. One of these methods is the virtual reality application, which has started to be used in the field of health with the developing technology, allowing individuals to experience another reality where they are. In addition, audio-visual (video) therapy methods are other methods that can be used in the symptom management of these patients. It is stated that virtual reality intervention and audio-visual therapies (relaxant video application) have positive effects on cancer patients and patients receiving chemotherapy treatment. In this study, the effect of interactive/immersive virtual reality intervention and relaxant video application on symptom severity, distress level and quality of life of patients diagnosed with lung cancer will be evaluated. Patients diagnosed with lung cancer, receiving chemotherapy treatment for the first time, and whose protocols are Cisplatine+Etoposide, Carboplatin+Etoposide, Paclitaxel+Carboplatine, Dosataxel+Cisplatine, Cisplatine+Pemetreksed, Carboplatine+Pemetreksed, Cisplatine+Vinorelbine, Gemsitebine+Cisplatine/Carboplatine and only Cisplatine, will be included in the study. Patients will be assigned to 3 groups: virtual reality application group (VR), relaxant video application group (RV) and control group (CG) by stratified randomization according to the disease stage and drug type. During the chemotherapy treatment, an interactive/immersive virtual reality intervention (VR group) and relaxant video intervention (RV group) consisting of nature-themed scenarios, which are preferred due to their relaxing effects, will be carried out for 2 times, about 20 minutes, the first day of each chemotherapy cycle, during 2 chemotherapy cycles. The control group will receive routine/standard nursing care. Research data will be collected at different intervals during the chemotherapy cures with the Patient Information Form (only once), the Edmonton Symptom Diagnosis Scale, the NCCN Distress Thermometer, the European Cancer Treatment and Organization Committee Quality of Life Scale and the Patient Follow-up Form and will be analyzed with the IBM SPSS v.23 program.

ELIGIBILITY:
Inclusion Criteria:

* are over 18 years old,
* diagnosed with lung cancer,
* will receive chemotherapy for the first time,
* will receive at least 2 cycles of chemotherapy treatment
* agree to participate in the study,

Exclusion Criteria:

* Having a cognitive and psychiatric disorder and diagnosis,
* Having brain metastasis or chronic disease related to the head-brain region,
* Having vision-hearing problems,
* Having epilepsy, vertigo, chronic severe headache, dizziness problems,
* Having a history of virtual reality, simulator or motion sickness,
* Having/declaring that he/she has open area, underwater, specific animal phobia,
* Do not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Edmonton Symptom Assessment Scale (ESAS) | First day of each chemotherapy cycle (totally 2 cycles) (2 times in about 21 days, totally 4 times in about 42 days or more)
  Changes on overall score of Edmonton Symptom Assessment Scale.
  The scale is a numerical scale between 0 and 10 developed to measure each symptom level (total 12 symptoms). Lower scores indicate lower symptom levels.

SECONDARY OUTCOMES:
National Comprehensive Cancer Network Distress Thermometer (NCCN-DT) | (Before and after the interventios/for control groups same time -20 mins.-) First day of each chemotherapy cycle (totally 2 cycles) (2 times in about 21 days, totally 4 times in about 42 days or more)
  Changes on overall score of Distress Scale.
  The scale is a numerical scale between 0 and 10 developed to measure stress levels. Lower scores indicate lower stress levels.
The European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-30) | First day of each chemotherapy cycle (totally 2 cycles) (2 times in about 21 days, totally 4 times in about 42 days or more)
  Changes on overall score of Quality of Life Scale.
  The scale is a multi-dimesion scale including total 30 questios to measure quality of life level. Minimum score is 0, and maximum score is 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No